CLINICAL TRIAL: NCT01779518
Title: An Expanded Access Phase 2 Study of Sofosbuvir With Ribavirin and With or Without Pegylated Interferon for 24 Weeks in Subjects Who Have Undergone Liver Transplantation and Who Have Aggressive, Recurrent Hepatitis C Infection
Brief Title: Expanded Access Program of Sofosbuvir With Ribavirin and With or Without Pegylated Interferon in Aggressive Post-transplant Hepatitis C
Status: Approved for marketing | Type: Expanded Access
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: GS-US-334-0139
Record Dates: First submitted 2013-01-23; First posted 2013-01-30 (Estimated); Last update posted 2014-01-16 (Estimated); Status verified 2014-01

CONDITIONS: Post-transplant Hepatitis C
Keywords: HCV; Sustained Virologic Response; Direct Acting Antiviral; GS-7977; Pegylated interferon; Ribavirin; Open Label; Sofosbuvir; Liver transplant; Hepatitis; Hepatitis, Chronic; Hepatitis C; Hepatitis C, Chronic; Liver Diseases; Digestive System Diseases; Hepatitis, Viral, Human; Virus Diseases; Enterovirus Infections; Picornaviridae Infections; RNA Virus Infections; Flaviviridae Infections; Antiviral Agents; Anti-Infective Agents; Therapeutic Uses; Pharmacologic Actions; Antimetabolites; Molecular Mechanisms of Pharmacological Action
MeSH Terms: conditions — Hepatitis; Hepatitis, Chronic; Hepatitis C; Hepatitis C, Chronic; Liver Diseases; Digestive System Diseases; Hepatitis, Viral, Human; Virus Diseases; Enterovirus Infections; Picornaviridae Infections; RNA Virus Infections; Flaviviridae Infections | interventions — Sofosbuvir; Ribavirin

INTERVENTIONS:
Drug: Sofosbuvir
  Other Names: GS-7977; PSI-7977; Sovaldi™
Drug: Ribavirin
Drug: Pegylated Interferon

SUMMARY:
This is a single arm, open-label study which will be opened at specific clinical sites at the request of an investigator for the treatment of individual subjects for whom there are no other treatment options. Subjects will be treated for 24 weeks with sofosbuvir (400mg QD) with RBV; pegylated interferon may be added at the discretion of the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Age > or = 18 years
* Previously undergone orthotopic liver transplant (OLT) at least 2 months prior to the planned start of dosing
* Aggressive Hepatitis C infection (including fibrosing cholestatic hepatitis C)
* Life expectancy of < 12 months if the HCV is left untreated

Exclusion Criteria:

* History of clinically significant drug allergy to nucleoside/nucleotide analogs
* Participation in a clinical study with an investigational drug or biologic within 1 month prior to anticipated dose administration, unless information is available to determine that there is no safety or drug-drug interaction risk to the subject
* Unable or unwilling to follow the contraception requirements

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult